CLINICAL TRIAL: NCT02187822
Title: A Phase 1 Study of TPI 287 Concurrent With Fractionated Stereotactic Radiotherapy (FSRT) in Treatment of Brain Metastases From Advanced Breast and Non-Small Cell Lung (NSCL) Cancer
Brief Title: Fractionated Stereotactic Radiotherapy (FSRT) in Treatment of Brain Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding by company providing TPI-287
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17816
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Brain Metastases; Generalized Malignancy, Primary; Brain Lesions
Keywords: Brain; Advanced solid tumors; Fractionated Stereotactic Radiotherapy (FSRT); Brain lesions; Primary solid malignancy
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — TPI-287; taxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation + Dose Expansion (Experimental): Dose Escalation followed by Dose Expansion.
  Dose Escalation Phase: The maximum tolerated dose (MTD) for TPI 287 given concurrently with Fractionated Stereotactic Radiotherapy (FSRT) will be determined using the standard 3+3 study design.
  Dose Expansion Phase: Participants will be treated with TPI 287 at MTD given concurrently with FSRT to further assess toxicity and tumor response.
  Interventions: Drug: TPI 287; Procedure: Fractionated Stereotactic Radiotherapy (FSRT)

INTERVENTIONS:
Drug: TPI 287 — TPI 287 is an infusion given through veins. Dose escalation will begin at 14 mg/m^2/dose. Dose expansion will begin at the maximum tolerated dose (MTD).
  Other Names: taxane
Procedure: Fractionated Stereotactic Radiotherapy (FSRT) — The prescription dose will be 25 gray (Gy) in 5 daily fractions delivered to the planning target volume (PTV).

SUMMARY:
The main purpose of this study is to see whether addition of TPI 287 to FSRT is safe and tolerable. Researchers also want to find out if adding TPI 287 to FSRT can help with better controlling the growth of brain lesions in people with brain metastases from their cancer.

DETAILED DESCRIPTION:
Standard of care for treatment of patients with brain metastases, which are considered not surgically removable, is radiation therapy to the brain lesions. This treatment is called Fractionated Stereotactic Radiotherapy (FSRT) and is given without chemotherapy and usually over 5 days.

Researchers of this study want to find out if adding an investigational drug, called TPI 287, to standard radiation therapy (FSRT) can help people with brain metastases from cancer. TPI 287 is a drug that is being tested and is not approved for sale in the United States by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed non-central nervous system primary solid malignancy.
* Must have pathologically or radiologically confirmed metastatic disease in the brain.
* Potential participants with up to 3 brain metastases (symptomatic and non-symptomatic) can be treated on this study. Maximum diameter of each brain lesion should be ≤ 5 cm. Maximum tumor volume ≤ 120 cc.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%).
* Life expectancy of greater than 12 weeks.
* Patients requiring treatment with corticosteroids are eligible.
* Treatment with non-enzyme inducing anti-seizure medications is allowed.
* Must have normal organ and marrow function.
* Systemic chemotherapy washout period ≥ 7 days. For investigational dugs and monoclonal antibodies washout period ≥ 5x drug half-life. There are no limitations on number of prior treatment regimens.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of TPI 287 administration.
* Prior brain surgery or radiation is allowed as long as the metastatic lesion(s) to be targeted in this study has not previously been treated with radiation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy within 1 week (6 weeks for nitrosoureas or mitomycin C) or investigational therapies/monoclonal antibodies within 5 half-life of investigational compound or those who have adverse events which are greater than grade 1 and are due to agents administered more than 1 week earlier. Bisphosphonates, endocrine therapy, and trastuzumab are permitted without restriction.
* Are receiving any other investigational agents.
* Previous treatment of the target lesions with radiation therapy.
* Have previously been treated with whole brain radiation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TPI 287.
* Have brain metastases secondary to germ cell tumor or lymphoma malignancy.
* Women who are pregnant or nursing (lactating).
* Known contraindication to enhanced MRI and CT scan.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled seizure activity or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of TPI 287 | Up to 2 years
  MTD of TPI 287 given concurrently with Fractionated Stereotactic Radiotherapy (FSRT) to treat brain metastases from advanced solid tumors.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 5 years
  The percentage of participants with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents. Complete Response (CR): The tumor is no longer seen on two sequential MRI scans, and the patient is on no steroids or only adrenal-maintenance dose of steroids. Partial Response (PR): ≥ 50% decrease in the product of two diameters of target lesions on two sequential MRIs, taking as reference the baseline product of two diameters, provided that the patient has not had his/her dose of steroids increased since the last evaluation period. Stable Disease (SD): The scan shows no change, taking as reference the smallest product of diameters while on study. Patient should be receiving stable or decreasing doses of steroids.
Progression Free Survival (PFS) Rate | Up to 5 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Response Evaluation Criteria in Solid Tumors (RECIST v.1.0) definition of Progression follows. One or more of the following must occur: 20% or greater increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Solmaz Sahebjam, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT02187822/Prot_SAP_000.pdf